CLINICAL TRIAL: NCT02403544
Title: Image-Guided Radiation Therapy (IGRT) Associated With Concurrent Capecitabine and Oxaliplatin in the Treatment of Locally Advanced or Inoperable Hepatocellular Carcinoma (HCC): A Phase I Study
Brief Title: Phase I Study of Image-Guided Radiation Concurrent With Double-Agent Chemotherapy for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Jing Jin, M.D., Vice Chair of Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-048; 13-102/778 (Other: Ethics Committee of Cancer Institute and Hospital)
Record Dates: First submitted 2015-03-24; First posted 2015-03-31 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Clinical Trial, Phase I; Concurrent Chemoradiation; Oxaliplatin; Capecitabine; Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy, Image-Guided; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CCRT Arm (Experimental): Patients recruited will be treated by concurrent chemoradiotherapy with IGRT and two cytotoxic agents: capecitabine and oxaliplatin. Capecitabine will be taken orally twice a day, from D1 to D14 while oxaliplatin will be given intravenously on D1 and D8, every 21 days. The doses of the two drugs will be escalated alternatively in each level group. The radiation will be given by IGRT and the dose is between 45 to 54Gy, 1.8-3Gy per fraction.
  Interventions: Radiation: IGRT; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Radiation: IGRT — IGRT: 45 to 54Gy, 1.8-3Gy per fraction.
  Other Names: Image-guided radiation therapy
Drug: Capecitabine — Capecitabine: by oral, D1-14, every 21 days, 600mg/m2 bid per day in level 1, and then escalated every another dose level.
  Other Names: CCRT concurrent chemotherapy 1 capecitabine
Drug: Oxaliplatin — Oxaliplatin: intravenously, D1 and D8, every 21 days, 30mg/m2 per day in level 1, and then escalated every another dose level.
  Other Names: CCRT concurrent chemotherapy 2 oxaliplatin

SUMMARY:
This is a phase I study to evaluate the safety of concurrent chemoradiation combining radiotherapy (IGRT) with two cytotoxic agents, capecitabine and oxaliplatin in patients with advanced or inoperable hepatocellular carcinoma.

DETAILED DESCRIPTION:
In this phase I study, patients with advanced or inoperable hepatocellular carcinoma, or those failed other strategies will be recruited. The primary tumor and nearby metastatic nodes will be irradiated with Image-Guided Radiation Therapy (IGRT) mostly with conventional fractions. During the course, oral capecitabine and intravenous oxaliplatin will be given concurrently. The maximum tolerated dose (MTD) for the two drugs will be determined during escalation according to the occurrence of dose limiting toxicities (DLT).

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* KPS≥80.
* Life expectancy≥16 months.
* Histopathologically or clinically diagnosed HCC.
* Barcelona-Clinic Liver Cancer (BCLC) 0-C without distant metastasis.
* The primary tumor is unresectable, inoperable or failed in other previous therapies.
* Child-pugh≤6 (Child A), Indocyanine green retention rate at 15min <20%.
* HGb≥100g/L, WBC≥3×109/L, NEUT≥1.5×109/L, PLT≥75×109/L, Creatine≤1.5mg/dl (UNL), Bun≤30mg/dl, Alanine aminotransferase/Aspartate aminotransferase/Alkaline phosphatase≤2.5×UNL, TBil≤1.5×UNL, Prothrombin time≤1.5×UNL, INR≤1.5.
* No prior liver or upper abdomen radiation therapy.
* No previous history of allergic reaction attributed to fluorouracil or platinum drugs.
* Be conscious and could cooperate and comply with protocols for the study, such as simulation, smooth breathing and positioning for radiotherapy.
* Be ready to be followed up.
* Fulfill dosages requirement for targets and dose limits for organs at risk.
* The patient should be under anti-hepatitis-virus therapy if indicated.
* Sorafenib should be discontinued 7 days before the start of irradiation.
* Subjects informed of the diagnosis of advanced HCC who are fully informed about the content of the study by the investigator using the written consent form, and give written consent to participate in the study of their own free will.

Exclusion Criteria:

* KPS≤70.
* Existing distant metastasis.
* Child-Pugh≥7, Indocyanine green retention rate at 15min ≥20%.
* Primary tumor within the liver is not to be irradiated.
* Past liver transplantation.
* Complications of cirrhosis: active gastrointestinal bleeding, hepatic encephalopathy, refractory ascites, peritonitis, hepatorenal syndrome, hepatopulmonary syndrome.
* Upper gastrointestinal bleeding within 3 months.
* Any other carcinomas, except cured non-melanoma skin carcinoma, treated in-situ cervical cancer and ≤T1 bladder cancer.
* After planning optimization, the physician still consider risky to treat the patient with the plan or the benefit is negligible.
* Not conscious or can not cooperate or comply with the protocol for the study.
* Previous history of allergic reaction attributed to fluorouracil or platinum.
* Patients with serious comorbidities or uncontrolled medical conditions that the investigator feels might compromise study participation (including but not limited to: myocardial infarction, congestive heart failure (NYHA>2), unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled psychotic disorders, uncontrolled hypertension and cerebrovascular disease with previous stroke within 6 months, serious infections，positive HIV test, poorly controlled diabetes mellitus with fasting blood-glucose >8mmol/L or 2-hour postprandial blood glucose >11mmol/L within the past month).
* Thrombolytic therapy within 4 weeks, or any concurrent anti-coagulant therapy.
* Pregnant, nursing, or possibly pregnant women, or women desiring to become pregnant during the study period.
* Participation in any investigational study within 4 weeks preceding the start of study treatment.
* Other cases judged by the investigator to be ineligible for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) for capecitabine and oxaliplatin | up to four weeks after the end of the treatment.

SECONDARY OUTCOMES:
Dose Limiting Toxicity (DLT) | up to four weeks after the end of the treatment.
In field recurrence rate (LR) or local failure free survival (LFFS) | From the completion of CCRT to 6, 12, 24, 36 months afterward.
Intrahepatic failure rate or intrahepatic failure free survival (IHFFS) | From the completion of CCRT to 6, 12, 24, 36 months afterward.
Extrahepatic failure rate or extrahepatic failure free survival (EHFFS) | From the completion of CCRT to 6, 12, 24, 36 months afterward.
Overall survival | From the completion of CCRT to 6, 12, 24, 36 months afterward.
Tumor response rate including complete response and partial response rates | 1 month and 3 month from the end of CCRT

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, doctor, Study Director — Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China